CLINICAL TRIAL: NCT03556280
Title: Multi-Center Study of Sensory Stimulation to Improve Brain Function (Overture Study)
Brief Title: Multi-Center Study of Sensory Stimulation to Improve Brain Function
Acronym: Overture
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cognito Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CA-0005
Record Dates: First submitted 2018-05-22; First posted 2018-06-14 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer Disease; Cognitive Impairment; Mild Cognitive Impairment; Dementia Alzheimers; Dementia, Mild; Dementia, Alzheimer Type; Dementia of Alzheimer Type; Dementia; Cognitive Impairment, Mild; Cognitive Decline
Keywords: Dementia; Alzheimer's Disease; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment Group (Experimental): Will use the Active GammaSense Stimulation System.
  Interventions: Device: GammaSense Stimulation System (Active Settings)
- Control Group (Sham Comparator): Will use the Sham GammaSense Stimulation System.
  Interventions: Device: GammaSense Stimulation System (Sham Settings)

INTERVENTIONS:
Device: GammaSense Stimulation System (Active Settings) — Proprietary auditory and visual sensory stimulation device.
  Arms: Treatment Group
Device: GammaSense Stimulation System (Sham Settings) — Proprietary auditory and visual sensory stimulation device.
  Arms: Control Group

SUMMARY:
The Overture Study is a randomized, controlled, single-blind multi-center clinical trial using the GammaSense Stimulation system to study safety, tolerability, and efficacy in people with mild to moderate cognitive impairment.

DETAILED DESCRIPTION:
The Overture Study (CA-0005) is a Phase I/II randomized, controlled, single-blind multi-center clinical trial using the GammaSense Stimulation device to study safety, adherence rates and efficacy in subjects with mild to moderate cognitive impairment (MMSE 14-26) who are age 55 and older.

Subjects who pass screening will be randomized (ratio 2:1 Treatment to Control). Subjects and their caregivers will be blinded to their randomization group, as will key raters at each site. The device will be used for 60 minutes daily during the 6-month therapy phase, followed by a one month safety follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* >= 55 Years old
* MMSE 14-26
* Prodromal Alzheimer's Disease (AD), AD or Mild Cognitive Impairment (MCI) due to AD
* Participation of a caregiver

Exclusion Criteria:

* Profound hearing or visual impairment
* Seizure Disorder
* Use of memantine (Namenda or Namzaric)
* Implantable devices (non-MR compatible)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale- Cognitive Subscale (ADAS-Cog) | Quarterly over 6 months
  A widely accepted, validated measure of cognitive function in Alzheimer's Disease consisting of 14 questions that result in a score ranging from 0 to 90 with higher scores representing greater cognitive impairment

SECONDARY OUTCOMES:
Amyloid PET/CT | Quarterly over 6 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Brain Matters Research, Delray Beach, Florida
  - Brain Matters Research, Stuart, Florida
  - ActivMed Practices & Research, Inc, Methuen, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey

REFERENCES:
- [Derived] Carbonell F, Zijdenbos AP, Hempel E, Hajos M, Bedell BJ. A novel method for harmonization of PET image spatial resolution without phantoms. EJNMMI Phys. 2025 Mar 14;12(1):23. doi: 10.1186/s40658-025-00740-9. PMID 40082316
- [Derived] Hajos M, Boasso A, Hempel E, Shpokayte M, Konisky A, Seshagiri CV, Fomenko V, Kwan K, Nicodemus-Johnson J, Hendrix S, Vaughan B, Kern R, Megerian JT, Malchano Z. Safety, tolerability, and efficacy estimate of evoked gamma oscillation in mild to moderate Alzheimer's disease. Front Neurol. 2024 Mar 6;15:1343588. doi: 10.3389/fneur.2024.1343588. eCollection 2024. PMID 38515445
- [Derived] Cimenser A, Hempel E, Travers T, Strozewski N, Martin K, Malchano Z, Hajos M. Sensory-Evoked 40-Hz Gamma Oscillation Improves Sleep and Daily Living Activities in Alzheimer's Disease Patients. Front Syst Neurosci. 2021 Sep 24;15:746859. doi: 10.3389/fnsys.2021.746859. eCollection 2021. PMID 34630050